CLINICAL TRIAL: NCT00501267
Title: A Randomized, Repeat Dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of Solabegron (GW427353) in Combination With Oxybutynin in Healthy Adult Subjects.
Brief Title: A Study To Test The Interaction of Two Medications for Treatment of Overactive Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B3C109868
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Overactive Bladder
Keywords: solabegron,; oxybutynin,; healthy adults,; drug interaction
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — solabegron; oxybutynin

INTERVENTIONS:
Drug: solabegron and oxybutynin

SUMMARY:
The purpose of this study is to determine the effect of repeat doses of solabegron and oxybutynin when taken alone or together

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males & females ages 18-65;
* Body weight >50kg; BMI between 19-32;
* Signed and dated informed consent; QTc Interval <450 msec;

Exclusion Criteria:

* Resting blood pressure >140/90 mmHg or HR >100 at screening;
* History of drug allergy or other allergy which, in the opinion of the PI, contraindicates their participation;
* Positive urine drug, alcohol or serum pregnancy test at screening and prior to dosing;
* Positive HIV, Hepatitis B, C at screening; use of medications (except acetaminophen)or vitamins or herbal supplements within 7 days or 5 half lives prior to dosing and during study;
* history of urinary retention, gastric retention, and other sever gastrointestinal motility conditions, uncontrolled narrow-angle glaucoma or who are at risk for these conditions;
* history of chronic constipation and/or regular laxative use; donation of more than 500mL of blood within 56 days prior to dosing;
* clinically relevant abnormality identified during screening process or any medical condition or circumstance making the subject unsuitable for participation based on the Investigators assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Absorption rate of solabegron and oxybutynin | as measured by multiple blood draws after repeat dosing

SECONDARY OUTCOMES:
To assess bladder function | prior to dosing Session 1 and post dose for each session

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States